CLINICAL TRIAL: NCT01397045
Title: Fast Track Rehabilitation Following Video-assisted Lung Segmentectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theagenio Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Nikolaos Barbetakis, Head of Thoracic Surgery Department, Theagenio Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Theagenio Thoracic Surgery 1
Record Dates: First submitted 2011-07-14; First posted 2011-07-19 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Multiple Pulmonary Nodules
Keywords: Lung; Nodule; Rehabilitation; VATS; Thoracotomy
MeSH Terms: conditions — Multiple Pulmonary Nodules | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Video-assisted lung segmentectomy (Active Comparator): Patients undergoing VATS segmentectomy
  Interventions: Other: VATS
- Mini thoracotomy (Other): Patients undergoing lung segmentectomy through a mini thoracotomy
  Interventions: Procedure: Mini thoracotomy

INTERVENTIONS:
Other: VATS — Video-assisted lung segmentectomy
  Arms: Video-assisted lung segmentectomy
Procedure: Mini thoracotomy — Mini muscle sparing thoracotomy for lung segmentectomy
  Arms: Mini thoracotomy

SUMMARY:
Aim of this prospective randomized study is to assess the safety and efficacy of video-assisted lung segmentectomy (Group B) comparing with mini muscle-sparing thoracotomy (group A) during diagnostic process for pulmonary nodules.

ELIGIBILITY:
Inclusion Criteria:

* Patients with undiagnosed multiple pulmonary nodules

Exclusion Criteria:

* Centrally located lesions
* previous thoracotomy
* extensive lung consolidation, and inability to achieve one lung ventilation

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Duration of hospital stay | Participants will be followed till home discharge, an average of 2 weeks

SECONDARY OUTCOMES:
postoperative morbidity | Participants will be followed till home discharge, an average of 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Thoracic Surgery Department, Theagenio Cancer Hospital, Thessaloniki, Greece